CLINICAL TRIAL: NCT01648816
Title: Interaction Between Genetic Factors and Maternal Stressors During Pregnancy in the Risk of Postpartum Depression
Acronym: IGEDEPP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 10056; 2010-A01315-35 (Other Grant/Funding Number: ID-RCB)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- postpartum depression: caucasian mothers with postpartum depression
- control: caucasian mothers without depression

SUMMARY:
"The prevalence of postpartum depression (PPD) is approximately 13%. PPD is associated with a higher maternal morbidity and mortality, and also with pervasive effects on the emotional, cognitive and behavioral development of the infant.

Stressful life events, socio-demographic and obstetrical risk factors have been associated with the risk of PPD. Genetics risk factors of PPD have also been identified. We are presently studying for the first time how maternal stressors may interact with genetic factors to increase the risk of PPD (Gene x Environment interaction)".

DETAILED DESCRIPTION:
"The prevalence of postpartum depression (PPD) is approximately 13%. PPD is associated with a higher maternal morbidity and mortality, and also with pervasive effects on the emotional, cognitive and behavioral development of the infant.

Stressful life events, socio-demographic and obstetrical risk factors have been associated with the risk of PPD. Genetics risk factors of PPD have also been identified. We are presently studying for the first time how maternal stressors may interact with genetic factors to increase the risk of PPD (Gene x Environment interaction).

We want first to analyze the allelic association between SNPs of 5-HT, HPA and neurodevelopment genes and PPD with a case control association study We then analyse the interaction between maternal stressors during pregnancy and SNPS of our candidate genes (CRHR1, 5-HTT, TPH, BDNF, HMCN1).

3000 Caucasian mothers are included after pregnancy in 8 maternities and are evaluated at the inclusion, at 8 weeks and at 1 year with DIGS, FISC, EPDS and HAD, Stressful life events (Paykel). Blood are collected for all subjects for DNA extraction.

At week 8 and 1 year after pregnancy we search PPD with EDPS and DSM-IV criteria of depression".

ELIGIBILITY:
Inclusion Criteria:

* Caucasian mothers included after pregnancy (J0-J4)

Exclusion Criteria:

* Age <18 years old, schizophrenia or mental retardation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: causasian mothers after pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 3338 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2016-09-04 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Depressed subjects at week 8 after delivery (EPDS and DSM I-V criteria for depression) | 8 weeks after delivery
  Postnatal depression detected by a possible depression (EPDS score > 8) and then confirmed (if EPDS score > 8) by DIGS DSM-IV depression criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Dubertret, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Louis Mourier Hospital, Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tebeka S, Le Strat Y, Etain B, Ray M, Mullaert J, Dubertret C; IGEDEPP Study Group. Childhood Trauma and Perinatal Depression: Data From the IGEDEPP Cohort. J Clin Psychiatry. 2021 Sep 7;82(5):20m13664. doi: 10.4088/JCP.20m13664. PMID 34496464